CLINICAL TRIAL: NCT01763801
Title: P-max or P-submax? This is the Question! A Prospective Randomized Search of the Most Reliable ECG Landmark for a Long Term Central Venous Catheter.
Brief Title: Optimization of EKG Method for Long Term Central Venous Catheter Tip Placement
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Campus Bio-Medico University (Other)
Responsible Party: Principal Investigator, Massimiliano Carassiti, Professor, Campus Bio-Medico University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CaraPros
Record Dates: First submitted 2013-01-03; First posted 2013-01-09 (Estimated); Last update posted 2013-01-09 (Estimated); Status verified 2013-01

CONDITIONS: Vascular Access Complication
Keywords: chemo port; intravenous electrocardiographic guidance; P maximal wave; P submaximal wave; catheter tip

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- P-Max group (Active Comparator): Includes cases in which the catheter tip was considered correctly positioned when the Maximal P wave was obtained
  Interventions: Device: P-Max
- P-Submax group (Active Comparator): Includes cases in which the catheter tip was considered correctly positioned when the Submaximal P wave was obtained
  Interventions: Device: P-Submax

INTERVENTIONS:
Device: P-Max — tip placement in correspondence to the P-Max on the ECG
  Arms: P-Max group
Device: P-Submax — tip placement in correspondence to the P-Submax on the ECG
  Arms: P-Submax group

SUMMARY:
Intravenous electrocardiographic guidance (IVECG) is a safe, reliable and accurate technique to correctly position the catheter tip. The investigators sought to evaluate the superiority of the P-maximal (P-max) wave compared to the P-submaximal (P-submax) wave in obtaining a more correct, safer and longer lasting device placement, with a lower incidence of complications and secondary misplacement.

DETAILED DESCRIPTION:
This prospective randomized trial was designed to observe the placement of long term iv catheters obtained with the IVECG method. Patients were randomised into 2 groups: in group A the catheter tip was placed in correspondence to the P-max, in group B in correspondence to the P-submax. We followed up the tip position by measuring the variation of its distances from the tracheal carina on multiplanar reconstructions of volumetric CT scans taken within a month (T0) and a year (T1) from the port implant.

ELIGIBILITY:
Inclusion Criteria:

* indication to chemo port insertion
* ability to give informed consent

Exclusion Criteria:

* younger than 18
* inability to give consent
* atrial fibrillation or flutter
* pace-maker or implantable cardioverter-defibrillator

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 326 (Actual)
Dates: Start 2011-07; Primary Completion 2012-02 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Distance between tracheal carina and distal end of the catheter | up to 10 months

CONTACTS AND LOCATIONS:
Overall Officials: Massimiliano Carassiti, Professor, Principal Investigator — Campus Bio-Medico University; Paola Proscia, Doctor, Principal Investigator — Campus Bio-Medico University
Locations (1):
- University Hospital Campus BioMedico, Rome, Italy